CLINICAL TRIAL: NCT05751317
Title: Phenotypic and Genotypic Variations of Enterococcus Spp. Isolated From Patients With Hospital Acquired Infections in Sohag University Hospitals, Egypt
Brief Title: Phenotypic and Genotypic Variations of Enterococcus Spp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mai Gamal Abdel Naser Abbas Khalifa, principal investigator, Sohag University
Other Study IDs: Soh-Med-23-02-10
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Isolation of Enterococci From Samples; Demonstration of Enterococci Antibiotic Susceptibility; Detection of Strains Enterococci Produce Biofilm; Studying Effect of Nanoparticles on Enterococci Antimicrobial Resistance; Studying Effect of Nanoparticles on Enterococci Biofilm; Genotyping of Enterococci
Keywords: phenotypic; genotypic; Enterococci; biofilm
MeSH Terms: interventions — Staining and Labeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Different samples (pus, urine, urinary catheter samples, stool, wound swabs, sputum, central venous catheter samples) will be collected under aseptic precautions from patients admitted at different departments at Sohag university hospitals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- samples containing Enterococci: Isolates of Enterococci will be identified by Gram staining, colony morphology, catalase test, and growth on Bile Esculin agar. All isolates will be identified to species level using Vitek2 automated system Strains confirmed as Enterococci will be examined for their antibiotic susceptibility by modified Kirby Bauer's disc diffusion method on MuellerHinton Agar.
  The biofilm formation activity of Enterococci isolates will be tested using the microtiter plate technique Detection of the effect of nanoparticles on the antibiotic susceptibility profile of Enterococci. Detection of the effect of nanoparticles on the biofilm producing Enterococci. Molecular identification of some virulence factors genes and antibiotic resistance genes of Enterococci using PCR
  Interventions: Diagnostic Test: Culture; Diagnostic Test: Staining:; Diagnostic Test: Biochemical reactions:; Diagnostic Test: VITEK; Diagnostic Test: Antibiotic sensitivity test; Diagnostic Test: nanoparticles effect; Diagnostic Test: The biofilm formation activity; Diagnostic Test: molecular diagnosis
- samples with bacteria other than enterococci
  Interventions: Diagnostic Test: Culture; Diagnostic Test: Staining:; Diagnostic Test: Biochemical reactions:; Diagnostic Test: VITEK

INTERVENTIONS:
Diagnostic Test: Culture — * Samples will be transported to Medical Microbiology and Immunology Laboratory and will be inoculated on MacConkey medium.
  * Pink colonies will be inoculated on bile esculin agar medium.
  * Enterococci produce blackening of the agar
Diagnostic Test: Staining: — The growing colonies on bile esculin agar medium will be examined microscopically after staining by Gram stain.
Diagnostic Test: Biochemical reactions: — * Catalase test.
  * Salt tolerance test
Diagnostic Test: VITEK — Automated identification of Enterococci will be done with VITEK2 system.
Diagnostic Test: Antibiotic sensitivity test — Strains confirmed as Enterococci will be examined for their antibiotic susceptibility by modified Kirby Bauer's disc diffusion method on Mueller-Hinton Agar.
  Groups: samples containing Enterococci
Diagnostic Test: nanoparticles effect — The effect of nanoparticles on Enterococci antimicrobial resistance pattern
  Groups: samples containing Enterococci
Diagnostic Test: The biofilm formation activity — The biofilm formation activity of Enterococci isolates will be tested using the microtiter plate technique
  Groups: samples containing Enterococci
Diagnostic Test: molecular diagnosis — Molecular identification of some virulence factors genes and antibiotic resistance genes of Enterococci using PCR
  Groups: samples containing Enterococci

SUMMARY:
Enterococci are Gram-positive facultative anaerobic cocci arranged in short and medium chains. Enterococci reside in the gastrointestinal tract and usually function commensally with humans. They can, however, cause several infections, such as urinary tract infections (UTIs), intra-abdominal infection, bacteremia, or endocarditis.

Among many species identified, E. faecalis and E. faecium are the most common species capable of causing infection and posing a threat of antimicrobial resistance, with E. faecalis accounting for the majority of infections.

DETAILED DESCRIPTION:
Enterococci are Gram-positive facultative anaerobic cocci arranged in short and medium chains.

Enterococci reside in the gastrointestinal tract and usually function commensally with humans. They can, however, cause several infections, such as urinary tract infections (UTIs), intra-abdominal infection, bacteremia, or endocarditis.

Among many species identified, E. faecalis and E. faecium are the most common species capable of causing infection and posing a threat of antimicrobial resistance, with E. faecalis accounting for the majority of infections.

Pathogenic species of enterococci express many virulence factors such as adhesins, gelatinase, Enterococcus surface protein, aggregation substances and cytolysins along with biofilm formation. These factors enhance the ability of the pathogen to invade, attach and survive through the acquisition of nutrients in the host tissue. Their presence in drug resistant strains increases the severity of the infection

Enterococci are intrinsically resistant to antibiotics such as aminoglycosides and β-lactam-based antibiotics. Moderate resistance to aminoglycosides is due to the intrinsic low permeability of the enterococcal cell wall to the large aminoglycoside molecules and is more prevalent in E. faecium than E. faecalis. Intrinsic β-lactam resistance is due to the overexpression of penicillin-binding proteins with low affinity for β-lactams, which makes E. faecalis more resistant to penicillin than E. faecium

Moreover, enterococci can readily acquire resistance to antimicrobials, and vancomycin-resistant enterococci (VRE) are among the priority pathogens for which new antibiotics are needed.

In addition, biofilm formation is one of the strategies for the enterococci to evade the host's immune response and the inhibitory or killing effects of antibiotics.

This self-produced extracellular matrix also provides a suitable microenvironment for enterococci to grow and facilitates the transmission of mobile genetic elements (MGEs) between bacteria. Enterococcal biofilms have been implicated in indwelling device-related infections such as prosthetic valve endocarditis, prosthetic joint infections and catheter-related infections.

Biofilm forming bacteria show resistance to many antibiotics and immune response which results in treatment failure. Given the difficulty of treating and eradicating biofilm associated infections, there is an unmet need for therapeutic options other than antibiotics to prevent biofilm formation.

Nanoparticles are attracting attention given their very small size and various antibacterial properties. Nanoparticles can interact with bacteria per unit area, which can make the antibacterial activity of nanoparticles more powerful. Nanoparticles can also initiate several bactericidal pathways, such as disrupting the bacterial membrane and release of intracellular components, making it difficult for bacteria to become resistant.

ELIGIBILITY:
Inclusion Criteria:

* All patients suffering from infections that can be caused by Enterococci.

Exclusion Criteria:

* All patients suffering from infections that aren't caused by Enterococci

Ages: 1 Month to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All the selected patients will be subjected to complete history taking (personal, clinical, associated comorbidities, history of drug intake, and length of hospital stay before sampling).
  * Collected samples will be transported to the Medical Microbiology and Immunology research laboratory as soon as possible.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Isolation and identification of Enterococci from different clinical samples | from April 2023 to December 2023
  Isolation and identification of Enterococci from different clinical samples (pus, urine, urinary catheter samples, stool, wound swabs, sputum, central venous catheter samples) will be collected under aseptic precautions from patients admitted at different departments at Sohag university hospitals.
Demonstration of Enterococci antibiotic susceptibility profile | from April 2023 to December 2023
  Strains confirmed as Enterococci will be examined for their antibiotic susceptibility by modified Kirby Bauer's disc diffusion method on Mueller-Hinton Agar.
Detection of strains of Enterococci which produce biofilm | from April 2023 to December 2023
  The biofilm formation activity of Enterococci isolates will be tested using the microtiter plate technique
Studying the effect of nanoparticles on Enterococci antimicrobial resistance pattern | from April 2023 to December 2023
  Inhibition zones of all groups will be compared to detect the effect of nanoparticles on Enterococci antimicrobial resistance pattern.
Studying the effect of nanoparticles on Enterococci biofilm producing ability | from December 2023 to March 2024
  The effect of nanoparticles on Enterococci biofilm producing ability
Genotypic characterization of Enterococci. | rom December 2023 to March 2024
  Molecular identification of some virulence factors genes and antibiotic resistance genes of Enterococci using polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mona F Mohamed, professor, Study Chair — Sohag University; Wesam A Abu El wafa, Study Chair — Sohag University
Locations (1):
- Faculty Of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferguson DM, Talavera GN, Hernandez LA, Weisberg SB, Ambrose RF, Jay JA. Virulence Genes among Enterococcus faecalis and Enterococcus faecium Isolated from Coastal Beaches and Human and Nonhuman Sources in Southern California and Puerto Rico. J Pathog. 2016;2016:3437214. doi: 10.1155/2016/3437214. Epub 2016 Apr 10. PMID 27144029